CLINICAL TRIAL: NCT06400888
Title: a Prospective, Randomized, Open-Label, Clinical Trial Study Comparing the Efficacy and Safety for Needle-Free Subcutaneous Injector and Conventional Intramuscular Injection of Mecobalamin in Diabetes Peripheral Neuropathy
Brief Title: Needle-Free Subcutaneous Injector and Conventional Intramuscular Injection of Mecobalamin in Diabetes Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Yuanjin Zhang, Chief Physician of Department of Neurology, Peking University Third Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M2024117; HP2024-03-501004 (Other Grant/Funding Number: 2024 Haidian District Health and Wellness Development Research Incubation Program)
Record Dates: First submitted 2024-04-09; First posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Peripheral Neuropathy
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- needle free subcutaneous injector of mecobalamin (Active Comparator)
  Interventions: Other: needle-free subcutaneous injector for Mecbl
- intramuscular injection of Mecbl (Active Comparator)
  Interventions: Other: intramuscular injection of Mecbl

INTERVENTIONS:
Other: needle-free subcutaneous injector for Mecbl — needle-free subcutaneous injector for Mecbl
  Arms: needle free subcutaneous injector of mecobalamin
Other: intramuscular injection of Mecbl — intramuscular injection of Mecbl
  Arms: intramuscular injection of Mecbl

SUMMARY:
The evaluation for efficacy and safety of needle-free subcutaneous injector and conventional intramuscular injection of mecobalamin for diabetic neuropathy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, age 18-70 years.
2. Participants who have been diagnosed with type 1 or type 2 diabetes for at least 1 year.
3. Meet the diagnosis of peripheral neuropathy according to neuroelectrophysiological examination.
4. According to the researchers' clinical judgment, blood glucose has been optimally controlled. The blood glucose was kept as stable as possible during the study. HbA1c level≤9% prior to screening, the variety is at least less than 2% within the 3-months before enrollment.
5. No history of eye trauma or corneal laser treatment.
6. No history of keratopathy or other intraocular ophthalmic disease.
7. No history of wearing contact lenses.
8. Have not taken medicines that affect corneal metabolism.
9. Did not take Mecbl or α-lipoic acid therapy within 3 months before screening.
10. Women of child bearing age (e.g., non-operative birth control or pausimenia less than 1 year) must be negative in the gonadotropin pregnancy test (urine) screening and receive effective contraception during treatment.
11. Signs the informed consent.
12. Subjects are willing and able to comply with the study visit schedule, treatment plan, laboratory tests and other study procedures.

Exclusion Criteria:

1. Have been diagnosed with a malignant tumor in the past 2 years.
2. The presence of other neurological disorders that researchers believe perhaps affect the evaluation of DPN.
3. The presence of skin diseases in the affected skin areas may affect the evaluation of DPN and injection according to the researcher's judgment.
4. Amputation of the ends of fingers and toes.
5. Participated in any other trials involving a study or post-marketing drug within 30 days of screening.
6. Subjects with clinically significant or unstable diseases, such as but not limited to acute cardiovascular diseases, cerebrovascular diseases, liver diseases, kidney diseases, respiratory diseases, blood diseases, immune system diseases, inflammatory or rheumatic diseases, uncontrolled infections, symptomatic peripheral vascular diseases, untreated endocrine diseases, etc.
7. Had donated blood within 30 days of the study treatment commencement (if applicable); or preparative blood donors during the study or 30 days after the end of treatment.
8. The WBC < 4000 / mm^2, neutrophils count <1500/mm^2, platelet count <100×109 /mm^2.
9. Clinically significant abnormalities in 12-lead ECG.
10. Subjects received combining transcutaneous electrical nerve stimulation (TENS) or acupuncture.
11. A history of intolerance or allergy to Mecbl or similar chemical compound.
12. Current or history presence of alcohol and/or other substance abuse within the past 1 year.
13. Other severe acute or chronic medical or psychiatric conditions or laboratory abnormalities that, in the determination of the investigator, may increase the risk associated with participating in the trial or using Mecbl, or that may affect the interpretation of the study results, may render the subject unfit to participate in the trial.
14. Inability and/or unwillingness to understand and/or comply with the plan.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-05-30 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
concentration of plasma vitamin B12 | baseline, half an hour, first hour, second hour, 8 weeks
  The plasma vitamin B12, biomarker for effective active metabolite for neural repair.
corneal confocal microscopy parameter: inferior whorl length | baseline, 8 weeks
  The corneal nerve fiber length in inferior whorl area.
corneal confocal microscopy parameter: corneal nerve fiber length | baseline, 8 weeks
  The corneal nerve fiber length per frame.

SECONDARY OUTCOMES:
neurological function scales score: the modified Toronto clinical neuropathy score (mTCNS) | baseline, 8 weeks
  mTCNS is a valid and reliable scale for staging of mild to moderate diabetic sensorimotor polyneuropathy. Value of 3 or more is recommended for the diagnosis of peripheral neuropathy.
neurological function scales score: Norfolk Quality of Life Questionnaire - Diabetic Neuropathy (QOL-DN) | baseline, 8 weeks
  A patient-reported outcomes measure reflecting small fiber, physical functioning/large fiber neuropathy, autonomic nerve function, symptoms, and activities of daily living. Ranges from -4 to 136, higher score indicates worse QOL.
neurological function scales score: Neuropathy Impairment Score (NIS) | baseline, 8 weeks
  Clinician assessments about cranial nerves and limbs for muscle weakness, sensation loss, and decreased reflexes. ranges from 0 to 244. Higher NIS reflect greater neuropathic impairment.
neurological function scales score: Neuropathy Impairment Score of the lower limbs plus seven tests (NIS(LL)+7 tests) | baseline, 8 weeks
  Neuropathy impairment score of the lower limbs plus seven tests includes muscle weakness, sensation loss, and decreased reflexes. Ranges from 0 to 88. More NIS-LL scores indicate greater neuropathic impairment.
neurological function scales score: Polyneuropathy disability (PND) score | baseline, 8 weeks
  Polyneuropathy disability grades of walking. 0-IV grades were measured. More score is more severe impairment.
neurological function scales score: DNS score | baseline, 8 weeks
  Score items are unsteadiness of gait, burning or aching sensation, pricking sensation and numbness. A score of one or more denotes the presence of neuropathy.
neurological function scales score: NDS score | baseline, 8 weeks
  Evaluation of pinprick sensation, vibration sensation and temperature sensation. A total of 10 points was adopted. A score of 6 - 8 denotes the presence of moderate DPN, and a score of 9 - 10 denotes severe DPN.
neuroelectrophysiological parameter: NCV | baseline, 8 weeks
  Nerve conduction latency
neuroelectrophysiological parameter: NCV | baseline, 8 weeks
  Nerve conduction velocity
neuroelectrophysiological parameter: NCV | baseline, 8 weeks
  Nerve conduction wave amplitude
neuroelectrophysiological parameter: SSR | baseline, 8 weeks
  Velocity of sympathetic skin response
neuroelectrophysiological parameter: SSR | baseline, 8 weeks
  Amplitude of sympathetic skin response